CLINICAL TRIAL: NCT06301789
Title: Effect of Adding Magnesium Sulphate as an Adjuvant to Bupivacaine in Ultrasound-guided Quadratus Lumborum Block for Postoperative Analgesia in Lower Abdominal Cancer Surgeries.
Brief Title: Role of Magnesium Sulphate as an Adjuvant to Bupivacaine in U.S Guided Quadratus Lumborum Block in Lower Abdominal Cancer Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Martha Aweda Soliman, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Quadratus lumborum block
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: QLB in Lower Abdominal Cancer Surgeries as a Post Operative Analgesia

STUDY DESIGN:
Intervention Model Description: Effect of adding Mg sulphate as an adjuvant to bupivacaine for postoperative analgesia in cases of lower abdominal cancer surgeries
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): receive pre-emptive ultrasound-guided quadratus lumborum block with 25 mL of 0.25% bupivacaine on each side of the abdominal wall before induction of GA.
  Interventions: Drug: Effect of adding Mg sulfate as an adjuvant to bupivacain in U/S guided QLB for postoperative analgesia in lower abdominal cancer surgeries
- InterventionalGroup (Experimental): received pre-emptive ultrasound-guided quadratus lumborum block with 25 mL of 0.25% bupivacaine plus 2 ml of magnesium sulfate 10 % on each side of the abdominal wall before induction of GA.
  Interventions: Drug: Effect of adding Mg sulfate as an adjuvant to bupivacain in U/S guided QLB for postoperative analgesia in lower abdominal cancer surgeries

INTERVENTIONS:
Drug: Effect of adding Mg sulfate as an adjuvant to bupivacain in U/S guided QLB for postoperative analgesia in lower abdominal cancer surgeries — Bilateral ultrasound-guided transmuscular (anterior) quadratus lumborum block will be performed Each patient will be placed in the lateral position. the transducer will be placed in a transverse orientation on the flank just cranial to the iliac crest, then slide posteriorly to obtain an image of the quadratus lumborum muscle.echogenic needle will be inserted in-plane with the ultrasound beam in a posterior-to-anterior direction through the quadratus lumborum muscle until the ventral fascia of the muscle penetrated. At this point, the needle directed toward the fascial plan between the quadratus lumborum and the Psoas muscle; the correct position of the needle tip will be confirmed by injecting 3 mL of saline to separate the fascial layers at the lateral aspect of the quadratus lumborum muscle. Thereafter, the needle will be advanced more posteriorly between the quadratus muscle and psoas major muscle

SUMMARY:
The aim of this study is to assess the efficacy of Mg sulfate ( 10% ) as an adjuvant to Bupivacain ( 0.25 % ) in an U.S guided QLB for postoperative analgesia and postoperative Morphine consumption in lower abdominal cancer surgeries.

DETAILED DESCRIPTION:
It is vital to apply adequate postoperative analgesia following lower abdominal surgeries of cancer because Postoperative pain not only affects the patients' rest but also produces a series of pathological reactions. Postoperative analgesia, including regional anesthesia, is very important which not only provides effective postoperative analgesia but also reduces the need for postoperative opioids.In recent years, various ultrasound-guided regional anethetic techniques have been extensively used. One of them is Quadratus lumborum block which can provide postoperative analgesia of the segmental innervation from T6 to L1. In which the Local anesthetics can spread through the thoracolumbar fascia to the paravertebral space, thereby blocking part of the sympathetic nerves . Clinical studies have shown that compared with the current widely used transverse abdominal block, QLB provides longer analgesia and wider block levels when the same dose of local anesthetic is used unlike traditional trunk block, QLB cannot use the sense of falling during puncture and can only be performed under ultrasound guidance, which has the advantages of being real-time and dynamic. Ultrasound-guided nerve block provides more accurate positioning and benefits for patients with less injury. Magnesium sulfate plays an important role in the physiological function of the human body. A large number of studies have reported the safety and effectiveness of adding magnesium sulfate as an adjuvant in various regional anethetic techniques . Therefore, we designed a prospective randomized controlled trial to compare the analgesic efficacy of combining magnesium sulfate with bupivacaine in QLB.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 80 years old
2. Both gender
3. Weight from 55 to 85 kg
4. ASA groups 2 and 3
5. Lower abdominal cancer surgeries

Exclusion Criteria:

* 1. Patient refusal 2. True local anesthetic allergy 3. Coagulopathy 4. Local infection at the procedure site 5. Psychic patients 6. Patient on chronic opioid use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia | First 24 hrs postoperative
  Total morphine consumption during first 24hr postoperative

REFERENCES:
- [Background] Pelausa EO. Otolaryngology in Atlantic Canada: practitioners' perspectives. J Otolaryngol. 1999 Feb;28(1):31-6. PMID 10077781
- [Background] Mintz S, Anavi Y, Sabes WR. Peripheral ameloblastoma of the gingiva. A case report. J Periodontol. 1990 Oct;61(10):649-52. doi: 10.1902/jop.1990.61.10.649. PMID 2231232
- [Background] Smith BE, Suchak M, Siggins D, Challands J. Rectus sheath block for diagnostic laparoscopy. Anaesthesia. 1988 Nov;43(11):947-8. doi: 10.1111/j.1365-2044.1988.tb05658.x. PMID 2975148